CLINICAL TRIAL: NCT00742131
Title: A Phase 1 Dose Escalation Study of the Safety and Pharmacokinetics of GSK1363089 (Formerly XL880) Administered Orally to Subjects With Solid Tumors
Brief Title: A Dose Escalation Study of the Safety and Pharmacokinetics of GSK1363089 (Formerly XL880) Administered Orally to Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MET111647; NCT00105924 (obsolete NCT alias)
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Solid Tumours
Keywords: MET inhibitor; c-Met; XL880; GSK1363089; Solid Tumors
MeSH Terms: interventions — GSK 1363089

ARMS (1):
- Subjects receiving GSK1363089 (Experimental): Eligible subjects will receive GSK1363089 administered orally as a cinnamon-flavored liquid or as solid capsules with the starting dose for cohort 1 as 0.1 milligram/kilogram. Subjects in cohorts 1, 2, and 3A will receive GSK1363089 in the liquid formulation, while Cohorts 3B, 4, 5, 6, 7, and 8 will receive GSK1363089 in the solid capsule formulation.
  Interventions: Drug: GSK1363089

INTERVENTIONS:
Drug: GSK1363089 — GSK1363089 will be administered orally as a cinnamon-flavored liquid (250 milligrams of GSK1363089 in 50 milliliters liquid [5 milligrams/milliliter] or 1000 milligrams of GSK1363089 in 50 milliliters liquid [20 milligrams/milliliter]) or as solid capsules of 20, 100, and/or 200 milligrams.

SUMMARY:
This clinical study is being conducted at two sites to determine the optimum dose, safety, and tolerability of GSK1363089 treatment in adults with solid tumors. This study is no longer recruiting subjects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor which is metastatic or unresectable with no known effective treatment measures,
* ECOG performance status of </= 2.
* Adequate bone marrow reserve, hepatic, renal, and cardiovascular function,
* Negative pregnancy test.

Exclusion Criteria:

* Chemotherapy within 4-6 weeks of the start of treatment,
* Radiotherapy within 4 weeks of the start of treatment,
* Known brain metastasis,
* Uncontrolled medical disorder such as infection or cardiovascular disease,
* HIV positive,
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03-17 (Actual); Primary Completion 2008-05-13 (Actual); Study Completion 2011-08-29 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and to assess the safety and tolerability of GSK1363089 administered orally (up to twelve different doses) to subjects with solid tumors | 3 years

SECONDARY OUTCOMES:
To evaluate pharmacokinetic (PK) and pharmacodynamic parameters of GSK1363089, radiographically evaluate the effects of GSK1363089 on tumors, evaluate tumor response after repeat administration of GSK1363089 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Eder JP, Shapiro GI, Appleman LJ, Zhu AX, Miles D, Keer H, Cancilla B, Chu F, Hitchcock-Bryan S, Sherman L, McCallum S, Heath EI, Boerner SA, LoRusso PM. A phase I study of foretinib, a multi-targeted inhibitor of c-Met and vascular endothelial growth factor receptor 2. Clin Cancer Res. 2010 Jul 1;16(13):3507-16. doi: 10.1158/1078-0432.CCR-10-0574. Epub 2010 May 14. PMID 20472683
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study MET111647 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MET111647?search=study&study_ids=MET111647#rs
- Available data/document: Informed Consent Form: MET111647 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MET111647 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MET111647 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MET111647 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MET111647 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MET111647 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MET111647 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register